CLINICAL TRIAL: NCT02966444
Title: Hunger, Satiety, and Metabolic Responses to High-fat Meals of Varying Fatty Acid Composition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Texas Christian University (Other)
Responsible Party: Principal Investigator, Jada Stevenson, Assistant Professor, Texas Christian University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: CT2016JS1
Record Dates: First submitted 2016-11-08; First posted 2016-11-17 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Body Weight Changes
MeSH Terms: conditions — Body Weight Changes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- MUFA-rich HF Meal (Experimental): High-fat meal rich in monounsaturated fatty acids
  Interventions: Other: MUFA-rich HF Meal
- PUFA-rich HF Meal (Experimental): High-fat meal rich in polyunsaturated fatty acids
  Interventions: Other: PUFA-rich HF Meal
- SFA-rich HF Meal (Experimental): High-fat meal rich in saturated fatty acids
  Interventions: Other: SFA-rich HF Meal

INTERVENTIONS:
Other: MUFA-rich HF Meal
  Arms: MUFA-rich HF Meal
Other: PUFA-rich HF Meal
  Arms: PUFA-rich HF Meal
Other: SFA-rich HF Meal
  Arms: SFA-rich HF Meal

SUMMARY:
This study evaluates the effects of dietary fatty acid composition from high fat meals on markers of hunger, satiety and metabolism.

ELIGIBILITY:
Inclusion Criteria:

* BMI of >18.5-24.9kg/m2
* Woman
* 18-40yrs of age

Exclusion Criteria:

* Evidence of weight loss or gain exceeding 5% of their body weight within the past 3 months.
* Plans to lose weight or begin a weight loss program between initiation of study and final testing.
* Plans to begin an exercise program or change current exercise routines between initiation of study and final testing.
* Is on a medically prescribed diet
* Does not consume breakfast regularly
* Rate less than 80% of foods offered in the buffet at 50mm or more on the 100mm VAS as palatable
* Medications that could influence appetite or sensory function
* Reports of metabolic or endocrine disease, gastrointestinal disorders, or history of medical or surgical events that could affect fat digestion and hormone signaling.
* Any chronic disease including type II diabetes, hypothyroidism, hyperthyroidism, cardiovascular disease, and cancer
* Any supplements that a subject begins taking between initiation of study and final testing.
* Anyone who is currently pregnant, lactating, or planning on becoming pregnant before the conclusion of this study.
* Anyone who has allergies to any of the components of the liquid meals
* Anyone who has donated blood in the last 20 days

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Peptide-YY | 18 months

SECONDARY OUTCOMES:
Visual Analog Scale | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Jada L Stevenson, PhD, Principal Investigator — Texas Christian University
Locations (1):
- Texas Christian University, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No